CLINICAL TRIAL: NCT00093600
Title: A Phase IB, Open-Label Study to Determine the Safety and Pharmacokinetics of Twice Daily Oral Dosing of PKC412 Administered in Combinations Sequentially and Concomitantly With Daunorubicin and Cytarabine for Standard Induction Therapy, and High Dose Cytarabine for Consolidation in Patients With Acute Myeloid Leukemia (AML)
Brief Title: PKC412, Daunorubicin, and Cytarabine in Treating Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOVARTIS-CPKC412A2106; UCLA-0308139-01 (Other: UCLA); CDR0000389242 (Other: PDQ (Physician Data Query))
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2015-03

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); untreated adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Congenital Abnormalities | interventions — Cytarabine; Daunorubicin; midostaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PKC412 administered sequentially (Experimental): twice daily oral dosing of PKC412 administered sequentially
  Interventions: Drug: midostaurin
- PKC412 administered concomitantly (Experimental): PKC412 administered concomitantly with standard induction daunorubicin and cytarabine therapy followed by high-dose consolidation therapy with cytarabine
  Interventions: Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: midostaurin

INTERVENTIONS:
Drug: cytarabine
  Arms: PKC412 administered concomitantly
Drug: daunorubicin hydrochloride
  Arms: PKC412 administered concomitantly
Drug: midostaurin
  Other Names: PKC412

SUMMARY:
RATIONALE: PKC412 may stop the growth of cancer cells by blocking the enzymes necessary for their growth. It may also increase the effectiveness of daunorubicin and cytarabine by making cancer cells more sensitive to the drugs. Drugs used in chemotherapy, such as daunorubicin and cytarabine, work in different ways to stop cancer cells from dividing so they stop growing or die. Combining PKC412 with chemotherapy may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best way to give PKC412 when given either after or together with daunorubicin and cytarabine in treating patients with newly diagnosed acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and tolerability of PKC412 administered sequentially or concurrently with induction chemotherapy comprising daunorubicin and cytarabine followed by consolidation therapy comprising high-dose cytarabine in patients with newly diagnosed acute myeloid leukemia.
* Compare the pharmacokinetics of these regimens in these patients.

Secondary

* Determine the efficacy of these regimens, in terms of response rate, disease-free survival, and overall survival, in these patients.
* Correlate genetic variation in drug metabolism genes, leukemia genes, and drug target genes with response in patients treated with these regimens.

OUTLINE: This is an open-label, multicenter study. Patients are alternately assigned to 1 of 2 induction treatment groups.

* Induction therapy:

  * Group I (sequential therapy): Patients receive daunorubicin IV over 30 minutes on days 1-3, cytarabine IV continuously on days 1-7, and oral PKC412 twice daily on days 8-21 in the absence of disease progression or unacceptable toxicity.
  * Group II (concurrent therapy): Patients receive daunorubicin and cytarabine as in group I and oral PKC412 twice daily on days 1-7 and 15-21 in the absence of disease progression or unacceptable toxicity.

In both groups, patients are evaluated on day 28. Patients with persistent disease receive a second induction course comprising daunorubicin IV over 30 minutes on days 1 and 2, cytarabine IV continuously on days 1-5, and oral PKC412 on the same schedule as their assigned treatment group. Patients with a complete response after course 1 or course 2 proceed to consolidation therapy.

* Consolidation therapy: Patients in both groups receive high-dose cytarabine IV over 3 hours twice daily on days 1, 3, and 5 and oral PKC412 on the same schedule as their assigned treatment group. Treatment repeats every 28-42 days for 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of consolidation therapy, patients in both groups continue to receive PKC412 alone, according to their assigned treatment group, every 28-42 days for up to 3 years in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed acute myeloid leukemia (AML)

  * Newly diagnosed disease
* No history of or newly diagnosed myelodysplastic syndromes, history of myeloproliferative disease, or secondary AML
* No CNS malignancy

PATIENT CHARACTERISTICS:

Age

* 18 to 60

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* AST and ALT ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* No active viral hepatitis

Renal

* Creatinine ≤ 1.5 times ULN
* No chronic renal disease

Cardiovascular

* Ejection fraction ≥ 50% by MUGA or echocardiogram
* No congestive heart failure
* No myocardial infarction within the past 6 months
* No poorly controlled hypertension
* No other cardiovascular disease

Pulmonary

* No pulmonary infiltrate, including those suspected to be infectious

  * Patients with pulmonary infection whose clinical symptoms have resolved are eligible provided there are no residual pulmonary infiltrates on chest x-ray

Other

* No gastrointestinal impairment or disease that would preclude absorption of study drugs
* No uncontrolled diabetes
* No active uncontrolled infection
* No other disease, except carcinoma in situ, that would preclude study participation
* No other severe or uncontrolled medical condition that would preclude study participation
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 5 days since prior growth factors
* No concurrent biological response modifiers

Chemotherapy

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy except radiation castration
* No concurrent radiotherapy

Surgery

* More than 14 days since prior surgical procedure except central venous catheter placement or other minor procedure (e.g., skin biopsy)

Other

* More than 30 days since prior investigational agents
* No other concurrent anticancer agents
* No other concurrent investigational drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2004-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Complete Response (CR) rate | cycle 1, day 14, cycle day 21 - 28, end of each cycle
  cycle = between 28 days and 42 days in duration

SECONDARY OUTCOMES:
CR rate by FLT3 mutation and treatment arm | CR:cycle 1, day 14, cycle day 21 - 28, end of each cycle, FLT3: monthly
Overall survival by FLT3 mutation status | time of death of any cause(FLT# - minthly)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Investigative Site, MD, Study Director — Novartis Investigative Site
Locations (6):
- United States (4):
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Dana Faber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - MD Anderson Cancer Center/University of Texas, Houston, Texas
- Germany (2):
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Mainz

REFERENCES:
- [Result] Stone RM, Fischer T, Paquette R, Schiller G, Schiffer CA, Ehninger G, Cortes J, Kantarjian HM, DeAngelo DJ, Huntsman-Labed A, Dutreix C, del Corral A, Giles F. Phase IB study of the FLT3 kinase inhibitor midostaurin with chemotherapy in younger newly diagnosed adult patients with acute myeloid leukemia. Leukemia. 2012 Sep;26(9):2061-8. doi: 10.1038/leu.2012.115. Epub 2012 Apr 27. PMID 22627678
- See also: Results for CPKC412A2106 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=14505